CLINICAL TRIAL: NCT05575609
Title: Relation Between Anthropometric Measurements and Balance in Children With Type 1 Diabetes
Brief Title: Relation Between Anthropometric Measurements and Balance in Children With Type 1 Diabetes Relation Between Anthropometric Measurements and Balance in Children With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Mahmoud Abd-elmonem, Assist Prof. Physiacl therapy for pediatric department, faculty of physical therapy , Cairo university, Cairo University
Other Study IDs: diabetes
Record Dates: First submitted 2022-09-27; First posted 2022-10-12 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes mellitus; anthropometric measurements; balance; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: children with Diabetes Mellitus, Type 1 — assessment of Relation between anthropometric measurements and balance in children with type 1 diabetes

SUMMARY:
Type 1 diabetes mellitus is the most common chronic metabolic disorder in children. Diabetic children who take proper nutrition and good care attain normal growth status. Factors affecting growth in diabetic patients include gender, age at diagnosis, duration of disease, glycemic control, and puberty status. Moreover, diabetes mellitus has negative impact on vestibular system, affect proprioception and lower limb muscle fatigue resulting in reduced balance.

DETAILED DESCRIPTION:
Limited literature is available regarding the relation between anthropometric measurements and balance in children with diabetes mellitus. Therefore, the current study will be conducted to investigate the relation between anthropometric measurements (weight, height and body mass index) and balance in children with diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as controlled T1DM.
* Age ranges from 7 to 11 years.
* From both sexes.
* Duration of the disease 3 to < 5 years.
* Same socioeconomic level.

Exclusion Criteria:

* Other hormonal diseases (hypothyroidism or hyperthyroidism).
* Hereditary sensory and autonomic neuropathy
* Significant visual disorders.
* Subjects participating in regular sports activities.
* History of fracture or surgery in the lower extremities in the past 12 months.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with T1DM will be selected from Abu El-Rish Hospial, Cairo University. Sample size estimation will be carried out based on a pilot study to determine the recruited number of participants. Participants will be recruited according to the following criteria.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
balance | baseline assessment
  HUMAC balance system will be used to assess balance
weight anthropometric measurement | baseline assessment
  the anthropometric measurement will be conducted using universal weight scale
height anthropometric measurement | baseline assessment
  the anthropometric measurement will be conducted using universal height scale

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed E Mohamed, B.S.C, Principal Investigator — Cairo university, faculty of physical therapy; Asmaa O Sayed, Phd, Study Chair — Cairo university, faculty of physical therapy; SHaima A Mohamed, PhD, Study Director — Cairo University
Locations (1):
- Amira Mahmoud Abd-elmonem, Giza, Egypt